CLINICAL TRIAL: NCT02011854
Title: Acupuncture and Traditional Chinese Medicine Combined With Rehabilitation Therapy for Post-stroke Shoulder-hand Syndrome in Community Hospital: a Multicenter，Randomized，Controlled Trial
Brief Title: Acupuncture for Post-stroke Shoulder-hand Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zouqin Huang (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Zouqin Huang, Attending physician, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PW2013A-41
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Shoulder-hand Syndrome
Keywords: acupuncture，rehabilitation,Shoulder-hand Syndrome
MeSH Terms: conditions — Reflex Sympathetic Dystrophy | interventions — Rehabilitation; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture with rehabilitation (Experimental): Electric acupuncture,Chinese medicine,Chinese medicine cupping,rehabilitation,To treat five times a week,Total course is eight weeks
  Interventions: Device: rehabilitation; Device: Acupuncture
- rehabilitation (Other): rehabilitation,To treat five times a week,Total course is eight weeks
  Interventions: Device: rehabilitation

INTERVENTIONS:
Device: rehabilitation — rehabilitation,To treat five times a week,Total course is eight weeks
Device: Acupuncture
  Arms: Acupuncture with rehabilitation

SUMMARY:
Shoulder-hand syndrome，a common complication of stroke patient，which is an important factor of limb function recovery.This research aims to observe the effect and safety of Acupuncture and Traditional Chinese medicine Combined with Rehabilitation Therapy for Post-stroke Shoulder-hand Syndrome.Furthermore, the investigators will promote the treatment in community hospital.

ELIGIBILITY:
Inclusion Criteria:

- Ischemic stroke and shoulder hand syndrome,conscious,For 2 weeks to 6 months,Patients with I or Ⅱ period.

Exclusion Criteria:

- Disturbance of consciousness,With shoulder joint disease or muscle disease,Patients with shoulder hand syndrome Ⅲ period,Serious primary diseases such as heart,liver and kidney,Mental illness.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) method Visual analogue scale (VAS) method Visual analogue scale (VAS) | 4 weeks and 8 weeks after treatment
  To evaluate the pain in shoulder joint

SECONDARY OUTCOMES:
Fugl-Meyer scale | 4 weeks and 8 weeks after treatment
  To evaluate the limb movement function

OTHER OUTCOMES:
Barthel index (BI) | 4 weeks and 8 weeks after treatment
  To evaluate patient's ability in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Huang Zouqin, Dcctor, Study Director — Pudong New Area TCM Hospital
Locations (1):
- Pudong New Area TCM Hospital, Shanghai, Shanghai Municipality, China